CLINICAL TRIAL: NCT06810596
Title: Comparing Glycemic Control Efficacy Between The National Health System and Suez Canal University Protocols of Intravenous Insulin Infusion for Diabetic Adults in ICU
Brief Title: Comparing Efficacy Between Two Protocols of Intravenous Insulin Infusion for Diabetic Adults in ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Aiman Al-Touny, Lecturer of Anesthesia and Intensive Care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4960#
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-11

CONDITIONS: Glycemic Control; Critical Care; Diabetes Mellitus
Keywords: Glycemic Control; Insulin Infusion Protocol; Critically ill
MeSH Terms: conditions — Diabetes Mellitus; Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suez Canal University variable rate Protocol (Active Comparator): Variable rate intravenous insulin infusion will be administrated according to random blood glucose and adjusted body weight (ABW).
  ABW = IBW + 0.33x (actual body weight - IBW)
  If the RBS level is 80 - 200 mg/dl, the Insulin infusion rate = RBS/ 100, and for insulin-sensitive patients = RBS/150 If the RBS level is 201 - 250 mg/dl, the Insulin infusion rate = RBS/ 80, and for insulin-sensitive patients = RBS/80 If the RBS level is 251 - 300 mg/dl, the Insulin infusion rate = RBS/ 60, and for insulin-sensitive patients = RBS/60 If the RBS level > 300 mg/dl, the Insulin infusion rate = 0.1 ml /kg/h adjusted body weight (Max: 10 unit/h)
  Interventions: Procedure: Insulin infusion protocol
- NHS group (Active Comparator): If the RBS level is 72- 144 mg/dl, the Insulin infusion rate = 1 ml/hr, for insulin-sensitive patients 0.5 ml/hr, and for Insulin resistance patients = 2 ml/hr If the RBS level is 145- 216mg/dl, the Insulin infusion rate = 2 ml/hr, for insulin-sensitive patients 1 ml/hr, and for Insulin resistance patients = 4 ml/hr If the RBS level is 217- 288 mg/dl, the Insulin infusion rate = 4 ml/hr, for insulin-sensitive patients 2 ml/hr, and for Insulin resistance patients = 6 ml/hr If the RBS level is 289- 360 mg/dl, the Insulin infusion rate = 5 ml/hr, for insulin-sensitive patients 3 ml/hr, and for Insulin resistance patients = 7 ml/hr If the RBS level is 361- 432 mg/dl, the Insulin infusion rate = 6 ml/hr, for insulin-sensitive patients 4 ml/hr, and for Insulin resistance patients = 8 ml/hr If the RBS level is >433 mg/dl, the Insulin infusion rate = 8 ml/hr, for insulin-sensitive patients 6 ml/hr, and for Insulin resistance patients = 10 ml/hr
  Interventions: Procedure: Insulin infusion protocol

INTERVENTIONS:
Procedure: Insulin infusion protocol — comparing the efficacy of 2 different protocols for glycemic control in diabetic critically ill patients.

SUMMARY:
The goal of clinical trial is to improve the adequacy of blood sugar control in diabetic critically ill adult patients who admitted to the intensive care unit(ICU) in Suez Canal University (SCU) hospitals by comparing glycemic control efficacy between the NHS in the UK and suggested SCU Protocols of Intravenous Insulin Infusion.

The main questions it aims to answer are:

Is SCU protocol of Intravenous Insulin Infusion more effective than NHS protocol in achieving blood glucose control targets in critically ill adult patients?

Researchers will compare glycemic control efficacy between the NHS in UK and suggested SCU Protocols of Intravenous Insulin Infusion for critically ill Adults in ICU to determine the best protocol in achieving good blood glucose control in diabetic critically ill adult patients in SCU Hospitals.

DETAILED DESCRIPTION:
Patients will be randomized into 2 equal groups; Group 1 (SCU group) will follow the SCU protocol of Intravenous Insulin Infusion in diabetic critically ill patients Group 2 (NHS group) will follow the NHS protocol of Intravenous Insulin Infusion in critically ill diabetic patients in UK.

Randomization will be done using a web randomizer and the randomization sequence will be concealed in numbered opaque envelopes that will be opened after patient enrollment to define his or her group assignment.

In both groups, control of blood glucose will be achieved with the use of an intravenous infusion of regular insulin in saline. Insulin will be administered, reduced, or discontinued according to the protocol in the different groups.

Two nurses must check and prepare the variable rate intravenous insulin infusion (VRIII) and every time the rate of infusion is changed. Insulin must be drawn up using an insulin syringe to draw up 50 units of prescribed Human Act rapid insulin and add to 49.5 ml of 0.9% sodium chloride in a 50 ml syringe. Mix thoroughly; this will provide a concentration of 1 unit / 1 ml.

VRIII will be stopped when RBS <80mg/dl and repeat the measure of RBS after one hour.

Laboratory investigations of routine blood tests will be requested on admission and at least once daily and in case of abnormal potassium level will be measured every 6 hours.

Regarding Serum K:

If K is 3.5-5.5 mmol/l- This is the target: total K+ given should be 1.5 mmol/kg/day If K is >5.5 mmol/l - no K is to be added to the infusion fluid this day. If K is <3.5mmol/l - K+ given should be 2.0 mmol/kg/day. K+ replacement will be initiated if there are ECG changes of hypokalemia. If K is <2.5mmol/l - bolus K+ replacement 1 mEq/kg will be infused over 3 hours and serum K+ level rechecked 2 hours after the end of infusion. If recheck serum K+ level < 2.5mmol/l bolus K+ replacement will be infused again over 3 hours. If recheck serum K+ level >3mmol/l K+ maintenance will be infused 2.0 mmol/kg/day.

Data collection :

At baseline, demographic and clinical characteristics, including the Acute Physiology and Chronic Health Evaluation II (APACHE II) score and the diagnostic criteria for severe sepsis will be collected.

Medical history :

1. Medical chronic disorders and the used treatment for them, such as hypertension, diabetes, liver or renal diseases .
2. Any known allergies to the drugs to be used . laboratory investigations:

a) Daily Routine Blood test (CBC, ABG, Electrolytes). b) Prothrombin time (PT), partial tissue thromboplastin time (PTT) and International randomized ratio (INR), Liver function tests and Kidney function tests every 3 days.

c) HBA1c on admission.

Follow up:

1. Nutrition: NPO, Enteral or parental.
2. Mechanical Ventilation days.
3. Complications: DKA, Hyperglycemia or Hypoglycemia.
4. ICU Discharge Date.
5. Hospital Discharge Date.

d) Outcome: Discharge or Death.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to the hospital with a potentially life-threatening condition (Critically ill patients) with HbA1C >6.0.

Exclusion Criteria:

* DKA patients.
* Pregnant or breast-feeding patients.
* Hyperosmolar Non-Ketotic Coma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Time needed to achieve the target blood glucose (80-180) | up to 28 days
  Assess the time needed to achieve the target blood glucose (80-180) in both protocols of intravenous insulin infusion in management of hyperglycemia in diabetic critically ill patients.

SECONDARY OUTCOMES:
Assess the effect of different factors in the management of hyperglycemia in critical ill patients. | up to 28 days
  Assess the effect of different factors in the management of hyperglycemia in critical ill patients (age, gender comorbidities, etc.)
Assess the incidence of hypoglycemia among the patients of both groups. | up to 28 days
  Assess the incidence of hypoglycemia among the patients of both groups.
Compare Ventilator Free Days between two groups. | up to 28 days
  Compare Ventilator Free Days between two groups
Compare the ICU stay and hospital stay between the two groups. | up to 28 days
  Compare the ICU stay and hospital stay between the two groups.
Compare ICU and 30 days Mortality rates between the two groups. | 30 days
  Compare ICU and 30 days Mortality rates between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University Hospitals, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication.
Access Criteria: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)